CLINICAL TRIAL: NCT04681287
Title: Exploratory Study of Advanced Breast Cancer in HER2 Positive Patients With Failure of Multi-line Therapy Treated by Combination of Inetetamab (Cipterbin) + PD-1 Inhibitor Combined With Utidelone.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-HER2-MBC001
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: HER2 Positive Metastatic Breast Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Patients with advanced HER2 positive breast cancer who had received at least paclitaxel, trastuzumab and TKIs (lapatinib or Pyrotinib) at least in the past were included in this study,Efficacy and safety of combination of inetetamab and PD-1 inhibitor combined with chemotherapy (including albumin bound paclitaxel, vinorelbine, gemcitabine, capecitabine or aribrin).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inetetamab and PD-1 inhibitor combined with chemotherapy. (Experimental)
  Interventions: Drug: inetetamab and PD-1 inhibitor combined with chemotherapy.

INTERVENTIONS:
Drug: inetetamab and PD-1 inhibitor combined with chemotherapy. — 1. Chemotherapy selected by doctors: albumin bound paclitaxel, vinorelbine, gemcitabine, capecitabine, and aribrin were administered according to clinical routine;
  2. The first dose was 8 mg / kg, followed by 6 mg / kg, once every 3 weeks
  3. PD-1 inhibitor 200mg D1 every 3 weeks as a cycle Treatment to disease progression or toxicity intolerance, or death from any cause.
  The efficacy was evaluated every 2 cycles and adverse events were recorded. After 4-6 cycles of treatment, if the patient is intolerable to chemotherapy for any reason, the chemotherapy can be stopped and the combination of inistumab and PD-1 can be continued.

SUMMARY:
This study plans to explore the efficacy and safety of chemotherapy combined with inetetamab and PD-1 inhibitors in HER2 positive advanced breast cancer who failed to receive trastuzumab and TKIs, and explore the dominant population of dual antibody combination to further guide the precise and individualized treatment of advanced HER2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old female patients;
2. The results showed that HER-2 was positive at least once in patients with recurrent and metastatic breast cancer confirmed by pathology: HER-2 (+ + +) was confirmed by immunohistochemistry; if HER-2 (+ +), fish / CISH was required to confirm HER-2 amplification;
3. Previous treatment (including neoadjuvant, adjuvant and rescue therapy) received at least trastuzumab and TKIs;
4. It is allowed that the previous rescue chemotherapy does not exceed 3 lines, and must be disease progression before being included in the study; it is allowed to receive rescue endocrine therapy; chemotherapy allows to receive one of the chemotherapy of albumin binding paclitaxel, vinorelbine, gemcitabine, capecitabine and aribrin;
5. At least one target lesion can be defined according to RECIST 1.1, and the target lesion has not received radiotherapy (or other local treatment), unless it progresses after the treatment;
6. Before the study, chemotherapy and targeted therapy must be completed for at least 2 weeks, and endocrine therapy and antiangiogenic drug treatment for 1 week;
7. ECoG PS: 0-1 points;
8. The expected survival time was more than 3 months;
9. The function of the main organs is normal, that is to say, it meets the following standards:

1）Blood routine examination standard should meet (no blood transfusion and blood products within 14 days, not used G-CSF and other hematopoietic stimulating factors were corrected)

* Hb≥90g/L；

  ②ANC≥1.5×109/L；

  ③PLT≥75×109/L； 2）Biochemical examination should meet the following standards:
* TBIL<1.5×ULN；

  * Alt, AST < 2.5 × ULN, liver metastasis < 5 × ULN;

    * Bun and Cr ≤ 1 × ULN or creatinine clearance rate ≥ 50ml / min (Cockcroft Gault formula).

      10.Women of childbearing age must have a pregnancy test (serum) within 7 days before enrollment, and the results are negative, and they are willing to use appropriate contraceptive methods during the trial and within 8 weeks after the last administration of the trial drug; 11.The subjects volunteered to join the study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. Symptomatic, uncontrolled brain metastases or leptomeningeal metastases.However, patients with stable condition after local treatment for 4 weeks could be enrolled;
2. There was effusion in the third space which could not be controlled by drainage or air pressure;
3. Interstitial lung disease, non-infectious pneumonia, memory pneumonia, pulmonary fibrosis and other diseases;
4. Those who have a history of live attenuated vaccine vaccination in the 28 days before the first study medication or are expected to receive live attenuated vaccine in the study;
5. Other malignant tumors in the past 3 years, excluding cervical carcinoma in situ, basal cell carcinoma of skin or squamous cell carcinoma of skin;
6. Patients with hypertension who could not be reduced to normal range after antihypertensive drug treatment (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
7. Suffering from serious or uncontrollable diseases, including but not limited to:

1) Active viral infection, such as HIV, HBV active phase (HBsAg positive and HBV-DNA ≥ 103, hepatitis C antibody positive); 2) Previous severe cardiovascular diseases: uncontrollable hypertension; myocardial infarction, unstable arrhythmia, congestive heart failure, pericarditis, myocarditis, etc. in the first six and six patients; according to NYHA standard, grade III ~ IV cardiac insufficiency, or left ventricular ejection fraction (LVEF) < 50% according to NYHA standard; 8.Patients with a history of psychotropic substance abuse and unable to quit or with mental disorders; 9.According to the judgment of the researchers, there are other patients with accompanying diseases that seriously endanger the safety of patients or affect patients to complete the study; 10.Pregnant or lactating women; 11.The researchers think it is not suitable for the participants.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate at 3 months（PFS rate） | Estimated up to 3 months
  The rate of events from date of randomization until observation of disease progression or death from any cause at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lv H, Sun T, Ling X, Liu X, Yang J, Zhang M, Niu L, Chen S, Liu Z, Wang C, Sun H, Wang J, Zeng H, Zhao S, Guo L, Feng Y, Zhang Z, Xia Q, Qiu R, Yan M. Inetetamab plus camrelizumab and utidelone for pretreated HER2-positive advanced breast cancer: a prospective, single-arm, phase 2 study. BMC Med. 2026 Jan 27. doi: 10.1186/s12916-026-04643-z. Online ahead of print. PMID 41593669